

# STATISTICAL ANALYSIS PLAN

A Multi-Center, Phase 2, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% Novel Formulation) Compared to Vehicle in Subjects with Dry Eye Disease

| Sponsor: | Aldeyra Therapeutics, Inc. |
|------------------|----------------------------|
| Protocol Number: | ADX-102-DED-013 |
| Author: | |
| Date: | 30-DEC-2019 |

2.0

Version:



A Multi-Center, Phase 2, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% Novel Formulation) Compared to Vehicle in Subjects with Dry Eye Disease

Protocol Number:

ADX-102-DED-013

Version:

2.0

Date:

30-DEC-2019

Statistical Analysis Plan Approval

| | STREET, STREET | 10011 |
|---|---|---|
| 1 | | |
| 53 70 | | |
| Prepared by: | | |
| STATE OF THE PARTY | | |
| The second second | | |
| 55 | | |
| CONTRACTOR OF THE PARTY OF | | |
| Reviewed by: | | |
| WHILE COMPANY | | |
| 40.00 | | |
| 472 | | |
| 1900 | | |
| Approved by: | | |
| 35 | | |
| 7.0 | | |
| The second second | | |
| THE PERSON NAMED IN | | |
| Approved by: | | |
| Pro-coloraba de Cara | | |
| 3 | | |
| 1 | | |



A Multi-Center, Phase 2, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% Novel Formulation) Compared to Vehicle in Subjects with Dry Eye Disease

Protocol Number: ADX-102-DED-013

Version: 2.0

Date: 30-DEC-2019

## **Statistical Analysis Plan Approval**





## **Table of Contents**

| | Introduction | 7 |
|-----|------------------------------------------------|------------------|
| | Study Objectives | 7 |
| .1 | Primary Measures | 7 |
| .2 | Key Secondary Measures | 7 |
| .3 | Secondary Measures | 7 |
| .4 | Exploratory Measures | 8 |
| .5 | Safety Measures | 8 |
| .6 | Statistical Hypotheses | 9 |
| | Study Design and Procedures | 9 |
| .1 | General Study Design | 9 |
| .2 | Schedule of Visits and Assessments | 10 |
| | Study Treatments | 13 |
| .1 | Method of Assigning Subjects to Treatment Arms | 13 |
| .2 | Masking and Unmasking | 13 |
| | Sample Size and Power Considerations | 14 |
| | Data Preparation | 14 |
| | Analysis Populations | 15 |
| .1 | Intent-to-Treat | 15 |
| .2 | Per Protocol | 15 |
| .3 | Safety | 15 |
| | General Statistical Considerations | 15 |
| .1 | Unit of Analysis | 15 |
| .2 | Missing or Inconclusive Data Handling | 16 |
| .3 | Definition of Baseline | 16 |
| .4 | Data Analysis Conventions | 16 |
| .5 | Adjustments for Multiplicity | 17 |
| | Disposition of Subjects | 17 |
| | Demographic and Pretreatment Variables | 18 |
| 0.1 | Demographic Variables | 18 |
| 0.2 | Pretreatment Variables | 18 |
| | Medical History and Concomitant Medications | 18 |
| 1.1 | Medical History | 18 |
| 1.2 | Concomitant Medications | 19 |
| | Dosing Compliance and Treatment Exposure | 19 |
| | 2 3 4 5 6 1 2 1 2 3 1 2 3 4 5 0.1 0.2 1.1 | Study Objectives |



| | 12.1 Dosing | g Compliance | 19 |
|---|---|---|---|
| | 12.2 Treatn | nent Exposure | 20 |
| 13 | . Efficac | y Analyses | 20 |
| | 13.1 Primar | y Analysis | 20 |
| | 13.1.1 | Ocular Dryness Score | 21 |
| | 13.2 Key Se | econdary Analysis | 22 |
| | 13.2.1 | Fluorescein Nasal Staining | 23 |
| | 13.3 Secon | dary Analyses | |
| | 13.3.1 | Fluorescein Nasal Staining | 25 |
| | 13.3.2 | Dryness from the Ora Calibra® Ocular Discomfort & 4-Symptom Questionna | ire25 |
| | 13.3.3 | Fluorescein Staining (Ora Calibra® Scale) | 26 |
| | 13.3.4 | Ocular Dryness (VAS) | 27 |
| | 13.3.5 | Ocular Dryness Score | 28 |
| | 13.3.6 | Fluorescein Nasal Staining | |
| | | | 28 |
| | 13.3.7 | Fluorescein Nasal Staining | 29 |
| | 13.3.8 | Dryness from the Ora Calibra® Ocular Discomfort & 4-Symptom Questionna | |
| | 10.0.0 | September 1 Star Sansta Second 1 Symptom Questioning | |
| 14 | . Explor | atory Analyses | 30 |
| | 14.1.1 | Visual Analog Scale | 31 |
| | 14.1.2 | Ocular Discomfort Scale (Ora Calibra Scale) | 32 |
| | 14.1.3 | Ocular Discomfort & 4-Symptom Questionnaire (Ora Calibra® Scale) | 32 |
| | 14.1.4 | Ocular Surface Disease Index <sup>©</sup> | 33 |
| | 14.1.5 | Symptom Assessment in Dry Eye | 35 |
| | 14.1.6 | Conjunctival Allergen Challenge Ocular Itching Scale (Ora Calibra® Scale) | 35 |
| | 14.1.7 | Lissamine Green Staining (Ora Calibra® Scale) | 36 |
| | 14.1.8 | Tear Film Break-Up Time | 37 |
| | 14.1.9 | Tear Osmolarity | 38 |
| | 14.1.10 | Unanesthetized Schirmer's Test | 38 |
| 15 | . Safety | Analyses | 39 |
| | 15.1 Advers | se Events | 39 |
| | 15.2 Visual | Acuity (ETDRS) | 41 |
| | 15.3 Slit-La | mp Biomicroscopy Examination | 41 |
| | 15 / Introo | cular Pressure | 12 |
| | 15.4 11111 400 | and 1 1000d10 | 72 |
| | | f Fundoscopy Examination | |



| 16. | Changes from Protocol-Stated Analyses | 43 |
|-----|---------------------------------------|----|
| 17. | Revision History | 43 |
| 18. | Tables | 44 |
| 19. | Listings | 49 |
| 20. | Figures | 51 |

## **List of Abbreviations**

| AE | Adverse Event |
|--------|-----------------------------------------------|
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| BID | Bis in die (Twice Daily) |
| CAC | Conjunctival Allergen Challenge |
| CAE | Controlled Adverse Environment |
| CI | Confidence Interval |
| CRO | Contract Research Organization |
| CS | Clinically Significant |
| eCRF | Electronic Case Report Form |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| FSN | Fluorescein Staining of the Nasal Region |
| ICH | International Conference on Harmonisation |
| IOP | Intraocular Pressure |
| IP | Investigational Product |
| ITT | Intent-to-Treat |
| ITTFSN | Intent-to-Treat Fluorescein Nasal Score |
| ITTOD | Intent-to-Treat Ocular Dryness |
| IWRS | Interactive Web Response System |
| logMAR | Logarithm of the Minimum Angle of Resolution |
| LS | Least Squares |
| MAR | Missing at Random |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mmHg | Millimeters of Mercury |
| MMRM | Mixed Model for Repeated Measures |
| MNAR | Missing Not at Random |
| mOsm | Milliosmoles |
| NCS | Not Clinically Significant |
| OD | Oculus Dexter (Right Eye) |
| OS | Oculus Sinister (Left Eye) |
| OSDI | Ocular Surface Disease Index |



| OU | Oculus Uterque (Both Eyes) |
|---------|---------------------------------------------|
| PDF | Portable Document Format |
| PP | Per Protocol |
| PPOD | Per Protocol Ocular Dryness |
| PPFSN | Per Protocol Fluorescein Nasal Score |
| PT | Preferred Term |
| QID | Quater in Die (Four Times Daily) |
| RTF | Rich Text Format |
| SAE | Serious Adverse Event |
| SANDE | Symptom Assessment in Dry Eye |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| SDC | Statistics & Data Corporation, Incorporated |
| SE | Standard Error |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TEAE | Treatment-Emergent Adverse Event |
| TFBUT | Tear Film Break-Up Time |
| TMF | Trial Master File |
| VA | Visual Acuity |
| VAS | Visual Analog Scale |
| WHODrug | World Health Organization Drug Dictionary |



#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and reporting for protocol ADX-102-DED-013, amendment 1 dated 17 December 2019.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline, entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, efficacy, and safety assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. The statistical analysis methods presented in this document will supersede the statistical analysis methods described in the clinical protocol. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the clinical study report.

### 2. Study Objectives

#### 2.1 Primary Measures

The primary efficacy measure for the trial are the following:

| • | | ocular dryness score measured by the |
|---|---------------------|--------------------------------------|
| | Visual Analog Scale | |





## 2.5 Safety Measures

The safety measures for the trial include the following:





| • | |
|---------|---------------------------------|
| i | |
| i | |
| 2.6 | Statistical Hypotheses |
| The fol | lowing hypothesis will be teste |

### 3. Study Design and Procedures

## 3.1 General Study Design

The clinical trial is a Phase 2, multicenter, randomized, double—masked, parallel-group, vehicle-controlled design with block enrollment. Subjects will be randomized to one of the following treatment groups at Visit 2 and will be instructed to follow a dosing regimen QID dosing for four weeks followed by BID dosing for weeks 5-12:

- Reproxalap Ophthalmic Solution (0.25% Novel Formulation)
- Vehicle Ophthalmic Solution (vehicle)

Approximately 200 subjects will be randomly assigned to one of the two treatment groups (1:1) to receive either Reproxalap Ophthalmic Solution (0.25% Novel Formulation) or vehicle solution as topical ophthalmic drops administered bilaterally QID for four weeks followed by BID dosing for weeks 5-12. Subjects, Sponsor, CRO and site personnel will be masked to treatment assignment.

During the screening period, two exposures to the CAE® will be conducted to ascertain eligibility to enter the study. Those who qualify will be randomized to receive study drug in a double-masked fashion for 84 days. Subjects will self-administer drops daily as instructed.



All subjects will dose with randomized treatment QID

The total number of expected participants, including screen failures, is approximately



Subjects who terminate early during the treatment period will be asked to complete safety assessments prior to commencement of alternative DED therapy (if possible). Subjects who are terminated early from the study will not be replaced.

Subjects, the Sponsor, the CRO, investigators, and site personnel will be masked to treatment assignment.

Table 1 shows the scheduled study visits, their planned study day (note that there is no Day 0 and that Day 1 corresponds to the day of randomization), and the acceptable visit window for each study visit:

Table 1. Scheduled Study Visits, Planned Study Days, and Visit Windows

| Scheduled Visit | Planned Study Day | Visit Window |
|-----------------|-------------------|--------------|
| Visit 1 | Day -14 | ± 2 Days |
| Visit 2 | Day 1 | N/A |
| Visit 3 | Day 8 | ± 2 Days |
| Visit 4 | Day 15 | ± 2 Days |
| Visit 5 | Day 29 | ± 2 Days |
| Visit 6 | Day 43 | ± 2 Days |
| Visit 7 | Day 57 | ± 3 Days |
| Visit 8 | Day 71 | ± 3 Days |
| Visit 9 | Day 85 | ± 3 Days |

#### 3.2 Schedule of Visits and Assessments

The schedule of visits and assessments is provided below for the study.



**Table 2. Schedule of Visits and Measurements** 









#### 4. Study Treatments

#### 4.1 Method of Assigning Subjects to Treatment Arms

Before the initiation of study run-in at Visit 1 (Day -14), each subject who provides written and informed consent will be assigned to a screening number. All screening numbers will be assigned in strict numerical sequence at a site and no numbers will be skipped or omitted. Each subject who meets all the inclusion and none of the exclusion criteria at Visit 1 (Day -14) and Visit 2 (Day 1) will be assigned a randomization number at the end of Visit 2 (Day 1). The Interactive Web Response System (IWRS) will be used to assign all randomization numbers.

| Ī |
|---|

Randomization and kit numbers will be assigned automatically to each subject as they are entered into the IWRS.

The site staff will dispense kit(s) required until the next visit. Both the randomization number and the dispensed study drug kit number(s) will be recorded on the subject's source document and electronic case report form (eCRF). The Sponsor, investigators, and study staff will be masked during the randomization process and throughout the study.

### 4.2 Masking and Unmasking

All subjects, investigators, and study personnel involved with the conduct of the study will be masked with regard to study drug treatment assignments. When medically necessary, the investigator may need to determine what treatment has been assigned to a subject. When possible (i.e., in non-emergent situations), Ora and/or the Sponsor should be notified before unmasking IP. Ora and/or the study Sponsor must be informed immediately about any unmasking event.

If an investigator identifies a medical need for unmasking the treatment assignment of a subject, he/she should contact Ora and/or the medical monitor prior to unmasking the identity of the IP, if possible. Ora will ask the site to complete and send them the Unmasking Request Form. Ora will notify Aldeyra and jointly will determine if the unmasking request should be granted. They may consult the medical monitor



as needed. The result of the request will be documented on the Unmasking Request Form. If approval is granted to unmask a subject, written permission via the Unmasking Request Form will be provided to the investigator. The investigator will unmask the subject using IWRS. The investigator will complete the Unmasking Memo form and include it in the subject's study file and provide a copy for the TMF (Trial Master File). For each unmasked request, the reason, date, signature, and name of the person who unmasked the subject, must be noted in the subject's study file.

Unmasked subjects will be discontinued from the study.

| 5. | Sample | Size | and | <b>Power</b> | Consider | ations |
|----|--------|------|-----|--------------|----------|--------|
|----|--------|------|-----|--------------|----------|--------|

| Based on the results of a Phase 2b clinical trial |
|---------------------------------------------------|

#### 6. Data Preparation

Electronic Case Report Forms (eCRF) will be developed by Statistics & Data Corporation, Incorporated (SDC). Unless otherwise specified by Aldeyra, the eCRFs will follow SDTM standards. Data from source documents will be entered into the eCRF by site personnel.

The clinical study database will be developed and tested in

After data are entered into the clinical study database, electronic edit checks and data review will be performed. All data validation specifications and procedures are detailed in the Data Validation Manual as a separate document. When the database has been declared to be complete and accurate, the database will be locked. Any changes to the database after data have been locked can only be made with the approval of Aldeyra and Ora in consultation with SDC.

All analyses outlined in this document will be carried out after the following have occurred:

| • |
|---|



| | • |
|------------|------------------------------------|
| 7. | Analysis Populations |
| 7.1 | |
| Inte | ent-to-Treat Population: |
| • | |
| _ | |
| 7.2 | Per Protocol |
| Per | -Protocol Population: |
| I | |
| _ | |
| 7.3 | Safety |
| <u>Saf</u> | ety Population: |
| 8. | General Statistical Considerations |
| 8.1 | Unit of Analysis |
| Saf | ety endpoints will be analyzed |



| 8.2 Missing or Inconclusive Data Handling |
|-----------------------------------------------------------------|
| The primary analyses using MMRM method will be performed |
| The printary analyses using william in mealed will be performed |
| 8.3 Definition of Baseline |
| Baseline measures are |
| 8.4 Data Analysis Conventions |
| All data analysis will be performed by SDC |



| 8.5 Adjustments for Multiplicity | |
|---------------------------------------|--------------|
| 9. Disposition of Subjects | |
| Subject disposition will be presented | |
| | اکس<br>البہا |



| | _ |
|-----------------------------------------------------|---|
| 10. Demographic and Pretreatment Variables | |
| 10.1 Demographic Variables | |
| The demographic variables collected | |
| | Ī |
| | _ |
| 10.2 Pretreatment Variables | |
| Baseline disease characteristics will be summarized | |
| | Ī |
| | į |
| | Ī |
| | _ |
| 11. Medical History and Concomitant Medications | |
| 11.1 Medical History | |
| Ocular medical history will be summarized | |
| | Ī |



| Listings of medical history will be generated separately for ocular and non-ocular data. |
|---|
| 11.2 Concomitant Medications |
| 11.2 Concomitant medications |
| Ocular and non-ocular concomitant medications will be coded |
| Listings of concomitant medications will be generated separately for ocular and non-ocular data. |
| 12. Dosing Compliance and Treatment Exposure |
| 12.1 Dosing Compliance |
| Dosing compliance |



| A subject listing of dosing compliance and study drug accountability will also be produced. |
|---|
| A subject listing of run-in, run-in instillation, and run-in replacement will be provided as well as study drug assignment, instillation, and replacement. |
| 12.2 Treatment Exposure |
| Extent of treatment exposure for completed or discontinued subjects will be calculated |
| Subject listings of study drug exposure and dosing compliance will be produced. |
| 13. Efficacy Analyses |
| 13.1 Primary Analysis The primary and point is |
| The primary endpoint is |



| The primary endpoint will be described in subject listings. |
|---------------------------------------------------------------------|
| <del></del> |
| 13.1.1 OCULAR DRYNESS SCORE |
| The subject will be asked to subjectively rate their ocular dryness |



| 13.2 Key Secondary Analysis |
|---|
| The key secondary endpoint is the overall mean change from baseline in fluorescein nasal region score |
| The key secondary endpoint will be described in subject listings |



### 13.2.1 FLUORESCEIN NASAL STAINING FROM WEEK 1 TO WEEK 6

| Scale |
|-------|



## 13.3 Secondary Analyses

| Secondary efficacy variables will be summarized |
|-------------------------------------------------|



| • |
|---|
| 13.3.1 FLUORESCEIN NASAL STAINING FROM WEEK 2 TO WEEK 12 |
| Fluorescein nasal staining will be graded using the Ora Calibra® Corneal and Conjunctival Staining |
| Scale |
| 13.3.2 Dryness from the Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire |
| Subjects will rate the severity of each of their symptoms |



| 13.3.3 FLUORESCEIN STAINING (ORA CALIBRA® SCALE) |
|--------------------------------------------------|
| Fluorescein staining will be conducted |



| 13.3.4 Ocular Dryness (VAS) through Visit 5 (Day 29) |
|------------------------------------------------------|
| Ocular dryness (OU) will recorded |



| 13.3.5 OCULAR DRYNESS SCORE | |
|-------------------------------------|---------|
| Ocular dryness score | will be |
| summarized | |
| 13.3.6 FLUORESCEIN NASAL STAINING | |
| Visit-based data will be summarized | |



| 13.3.7 FLUORESCEIN NASAL STAINING |
|---|
| Visit boood data will be a proposited |
| Visit-based data will be summarized |
| 13.3.8 DRYNESS FROM THE ORA CALIBRA® OCULAR DISCOMFORT & 4-SYMPTOM QUESTIONNAIRE |
| Visit bood data will be a preparited |
| Visit-based data will be summarized |



| 14. Exploratory Analyses |
|---------------------------------------------------|
| Exploratory efficacy variables will be summarized |



| • | |
|--------|-----------------------------------|
| i | |
| - | |
| _ | |
| Ī | |
| • | |
| | VISUAL ANALOG SCALE |
| Ocular | symptoms of the VAS will recorded |



| 4440. 0 |
|-------------------------------------------------------------------------|
| 14.1.2 OCULAR DISCOMFORT SCALE (ORA CALIBRA SCALE) |
| Ocular discomfort scores will be subjectively graded |
| 14.1.3 OCULAR DISCOMFORT & 4-SYMPTOM QUESTIONNAIRE (ORA CALIBRA® SCALE) |
| Subjects will rate the severity of each of the following symptoms |
| Carjoste IIII late the severity of each of the following symptoms |



| 14.1.4 OCULAR SURFACE DISEASE INDEX® |
|--------------------------------------|
| The OSDI <sup>®</sup> is assessed |





### 14.1.5 SYMPTOM ASSESSMENT IN DRY EYE

| Subjects will be asked to complete the SANDE Questionnaire |
|---|
| 14.1.6 CONJUNCTIVAL ALLERGEN CHALLENGE OCULAR ITCHING SCALE (ORA CALIBRA® SCALE) |
| Subjects will rate the severity of their ocular itching symptom |


| · |
|---|
| 14.1.7 LISSAMINE GREEN STAINING (ORA CALIBRA® SCALE) |
| 14.1.7 LISSAMINE GREEN STAINING (ORA CALIBRA® SCALE) Subjects will undergo lissamine green staining |



| 14.1.8 TEAR FILM BREAK-UP TIME |
|--------------------------------|
| The TFBUT will be recorded |



## 14.1.9 TEAR OSMOLARITY

| Tear osmolarity will be measured |
|--------------------------------------------------|
| 14.1.10 Unanesthetized Schirmer's Test |
| Unanesthetized Schirmer's test will be conducted |



| | | <br> | <br> |
|---|---|------|------|
| - | - | | |

### 15. Safety Analyses

All safety analyses will be conducted using the Safety population.

#### 15.1 Adverse Events

An AE is defined as any untoward medical occurrence associated with the use of an IP in humans, whether or not considered IP-related. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IP, without any judgment about causality. An AE can arise from any use of the IP (e.g., off-label use, use in combination with another drug or medical device) and from any route of administration, formulation, or dose, including an overdose.

All AEs will be coded using the MedDRA 22.0.

Treatment-emergent adverse events (TEAE) are defined as any event that occurs or worsens on or after the day that randomized study treatment is initiated. Adverse events recorded in the eCRF which began prior to treatment will not be included in the summary tables but will be included in the AE data listings.

An overall summary will be presented that includes the number and percentage of subjects who experienced at least one AEs, ocular AEs, non-ocular AEs, SAEs, AEs by maximal severity, AEs by relationship to study drug, AEs leading to treatment discontinuation, and AEs resulting in death by treatment arm for the Safety population. In addition, overall TEAEs and the number and percentage of subjects who experienced at least one TEAE, ocular TEAEs, non-ocular TEAEs, TE-SAEs, TEAEs by



maximal severity, TEAEs by relationship to study drug, TEAEs leading to treatment discontinuation, and TEAEs resulting in death by treatment arm for the Safety population.

Separate summaries will be provided for the following categories of AEs:

- Ocular AEs by SOC and PT
- Non-ocular AEs by SOC and PT
- Ocular TEAEs by SOC and PT
- Non-ocular TEAEs by SOC and PT
- Ocular TEAEs by SOC, PT, and maximal severity
- Non-ocular TEAEs by SOC, PT, and maximal severity
- Ocular TEAEs by SOC, PT, and strongest relationship to study drug
- Non-ocular TEAEs by SOC, PT, and strongest relationship to study drug
- Ocular TEAEs by SOC, PT, maximal severity, and strongest relationship to study drug
- Non-ocular TEAEs by SOC, PT, maximal severity, and strongest relationship to study drug
- TEAEs That Led to Premature Discontinuation
- SAEs

Adverse Events and TEAEs will be summarized using discrete summary statistics and presented by treatment arm and all subjects for the the Safety population. If a subject reports the same PT multiple times within the same SOC, that PT will only be reported once within that SOC. As with the PT, if a subject reports multiple conditions within the same SOC, that SOC will only be reported once. In the summary, SOC will be listed in ascending alphabetical order; PTs will be listed in order of descending frequency for all subjects within each SOC.

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the investigator or reported to him/her by the subject. The assessment of severity is made irrespective of relationship to IP or seriousness of the event and should be evaluated according to the following scale:

- Mild: Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate: Event is bothersome, possibly requiring additional therapy, and may interfere with the subject's daily activities.
- Severe: Event is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.

Subjects experiencing more than one AE within a given SOC or PT are counted once within that SOC or PT for the maximal severity.



The relationship of each AE to the study drug should be determined by the investigator using these explanations:

- Definitely Related: Relationship exists when the AE follows a reasonable sequence from the time of IP administration, follows a known response pattern of the drug class, is confirmed by improvement on stopping the IP and no other reasonable cause exists.
- Probably Related: Relationship exists when the AE follows a reasonable sequence from the time of IP administration, follows a known response pattern of the drug class, is confirmed by improvement on stopping the IP and the suspect IP is the most likely of all causes.
- Possibly Related: Relationship exists when the AE follows a reasonable sequence from the time
  of administration, but could also have been produced by the subject's clinical state or by other
  drugs administered to the subject.
- Unlikely to be related: Relationship between the AE and IP is more than likely to be unrelated
  to IP administration but the relationship cannot be definitely attributed to another cause.
- Not Related: Concurrent illness, concurrent medication, or other known cause is clearly
  responsible for the AE, the administration of the IP and the occurrence of the AE are not
  reasonably related in time, OR exposure to IP has not occurred.

Subjects experiencing more than one AE within a given SOC or PT are counted once within that SOC or PT for the maximum relationship. All AEs, ocular AEs, non-ocular AEs, and SAEs will be presented in subject listings.

# 15.2 Visual Acuity (ETDRS)

| The logarithm of the minimum angle of resolution (logMAR) VA | |
|--------------------------------------------------------------|---------|
| . A S | subject |
| listing of VA will also be produced. | |
| 15.3 Slit-Lamp Biomicroscopy Examination | |
| Slit lamp biomicroscopic observations will be graded | |



| parameters will also be produced. | A subject listing of the slit-lamp biomicroscopy |
|---|---|
| 15.4 Intraocular Pressure | |
| Intraocular pressure will be measured | |
| | A subject listing of IOP |
| will also be produced. | A subject listing of for |
| 15.5 Dilated Fundoscopy Examination | |
| Dilated fundus exams will be performed | |



| | A subject listing of the dilated fundoscopy |
|---|---|
| parameters will also be produced. | |
| 16. Changes from Protocol-Stated Analyses | |

17. Revision History



| Protocol ADX-102-DED-013 SAP, Version 2.0 | STATISTICS & DATA CORPORATION |
|-------------------------------------------|-------------------------------|













| 19. Listings | · |
|--------------|---|





